CLINICAL TRIAL: NCT04257981
Title: Effect of Transcranial Direct Current Stimulation Augmented With Activities in Virtual Reality on Functional Recovery of the Upper Extremity of Children With Hemiparesis
Brief Title: Effect of Transcranial Direct Current Stimulation on Upper Extremity of Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Collaborators: Shiekh Abdullah Al-Twejeri Research Chair for Stroke (Unknown)
Responsible Party: Principal Investigator, faizan kashoo, PT, Prinicipal investigator, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU/RBI/346754/1-3-2020
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-09

CONDITIONS: Cerebral Palsy Infantile
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Group 1: Transcranial direct stimulation + virtual related group: The group will receive the tCDS and VR Group 2: Sham Transcranial direct stimulation Group + virtual related group: The groups will only receive sham tCDS and VR.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Children will be randomly allocated to one of the two groups by the lottery method. The researcher involved in randomization will not be involved in the assessment or treatment of the participants. The participants and therapists will also be blinded about the subjects allocated to a group by assigning a unique random number to the participants. Pre and post assessment will be performed by the same therapist. The therapist involved in the treatment is blinded about the treatment received by other groups. Each participant will undergo 3 weeks of treatment, 4 days a week. The total number of treatment sessions for each participant will be 12. Each participant will be assessed on the baseline, 2nd week, 3rd week and on 8th week follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Transcranial direct stimulation + virtual related group:
  Brain stimulator v3.0 will be used to deliver 1.5 mA current over the scalp corresponding to the primary motor cortex. The current will be delivered via two surface electrodes 5 × 5 cm placed on the scalp Virtual reality (KVR) is the use of a computer interface involving upper limb activity in pediatric rehabilitation. VR creates an artificial environment, presented to the user through appropriate sensory stimulations.
  Interventions: Device: Brain stimulator v3.0
- Control group (Sham Comparator): Sham Transcranial direct stimulation Group + virtual related group; The sham set-up will follow a similar protocol as the experimental group but the intensity of the current will be ceased after 30 seconds of stimulation. Participants in the Sham group will feel the identical sensation as the experimental group and will be unable to differentiate between actual and sham tDCS such procedure is validated in earlier studies.
  Interventions: Other: Sham Comparator: Control group

INTERVENTIONS:
Device: Brain stimulator v3.0 — Brain stimulator v3.0 will be used to deliver 1.5 mA current over the scalp corresponding to the primary motor cortex. The current will be delivered via two surface electrodes 5 × 5 cm placed on the scalp, validated by the previous research
  Arms: Experimental group
Other: Sham Comparator: Control group — The sham set-up will follow a similar protocol as the experimental group but the intensity of the current will be ceased after 30 seconds of stimulation. Participants in the Sham group will feel the identical sensation as the experimental group and will be unable to differentiate between actual and sham tDCS such procedure is validated in earlier studies
  Arms: Control group

SUMMARY:
Purpose: The aim of the study is to determine the combined effect of transcranial direct current stimulation (tDCS) and activities in virtual reality on the functional recovery of the upper extremity function of the children with hemiparesis. Subjects: Forty children with infantile stroke with age group between (6-12 years) will be divided into two groups, the experimental group will receive tDCS plus VR while the control group will receive sham tDCS plus VR. All the children will receive tDCS for 30minutes with 1.5 mA intensity over the dominant motor cortex. Both groups will be treated for three times a week for 6 weeks. Instrumentation: The the Fugl-Meyer assessment, motricity index, and Modified Barthel index will be used to assess the dependent variables after the intervention.

DETAILED DESCRIPTION:
One in 4000 full-term infants develops arterial ischemic stroke at the time of birth.5 These children are commonly called an infantile stroke, infantile hemiplegia, perinatal stroke, and congenital hemiplegic cerebral palsy. Epileptic seizures are common in 24-45 % of children suffering from an infantile stroke within a month.6 Noninvasive brain stimulation (NIBS) is the novel method of delivering therapeutic currents to the brain for the purpose of diagnosis and treatment 7. There is an exponential increase in researches on the effect of NIBS on cognitive deficits. The NIBS has proven to cause neural modulation at the cortical level8. The effect of stimulation is either increased or decreased in neuronal activity, depending on the anodal and cathodal stimulation, firing rate, and period of the activation or inhibition910. There are two types of NIBS techniques safely practiced among humans, these are, Transcranial Magnetic Stimulation (TMS) and Transcranial Direct Current Stimulation (tCDS)11. tCMS uses a weak magnetic field that transforms into beneficial currents into the brain for diagnostic (Single-pulse tCMS) or treatment purposes (repetitive tCMS). The inhibitory or excitatory cortical effects are achieved by decreasing or increasing the frequency and duration of tCMS 12. tCDS involves the use of weak direct or alternating current applied on the scalp via electrodes for the purpose of neural modulation13. The most popular form of tCDS device is a battery-operated stimulator capable of producing direct current ranging from 0.5-2.0 mA14. Neural modulation is achieved by altering the resting membrane potential. The anode causes increased excitability due to its depolarizing effect whereas the cathode electrode causes inhibition due to the hyperpolarization effect14.

Virtual reality (KVR) is the use of a computer interface involving upper limb activity in pediatric rehabilitation. VR creates an artificial environment, presented to the user through appropriate sensory stimulations. Participants use the motion sensor mounted on the paretic hand to interact with the virtual environment. The participants will receive visual and auditory feedback. The purpose of the study is to evaluate the combined effect of virtual reality activities and tDCS on upper limb activity in children with hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

1. The congenital stroke survivors with mild to moderate degree of upper limb disability on the Brunnstrom recovery scale16. The scores from 3-4 are considered moderate and 5-6 as a mild degree of upper-limb disability.
2. Age 5-12 years.
3. Able to understand simple commands.
4. Normal vision or with corrected glass

Exclusion Criteria:

1. Hemorrhage in the subarachnoid space
2. Aphasia
3. Neurosurgery of brain
4. Seizures in the past 12 months.
5. On medication for seizures.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Baseline and post- intervention Fugl-Meyer motor assessment | 8 Months
  The Fugl-Meyer motor assessment (FM) will be the primary outcome measure. The scale is a reliable and valid measure for upper limb impairment among stroke patients19. The score ranges from 0-66, score less than 18 are considered severe to moderate functional impairment. The scale takes 20 minutes to complete.

SECONDARY OUTCOMES:
Beiseline and post- intervention Motricity Index | 8 Months
  : Motricity Index (MI) upper limb items will be used to evaluate upper limb strength. The tool is found valid and reliable20 in scoring upper limb strength in stroke patients.
Baseline and post- intervention Modified Barthel Index | 8 Months
  Modified Barthel Index (BI) is a valid tool21 to measure functional disability in neurological disability to evaluate the functional disability. The scale will take 45 minutes to administer.

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Faizan Kashoo, Riyadh, Riyadh Region
  - Faizan Kashoo, Riyadh

IPD SHARING:
Plan to Share IPD: No
Data will be shared by the authors upon request.